CLINICAL TRIAL: NCT07298135
Title: A Randomized, Open-Label, Controlled Study to Evaluate the Effects of a Prebiotic Soda on Glycemic Control in Adults With Glucose Dysregulation
Brief Title: A Study to Evaluate the Effects of a Prebiotic Soda on Glycemic Control in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olipop, PBC (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20254308
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Blood Glucose Control

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be randomized to replace traditional non-diet soda with prebiotic soda
  Interventions: Behavioral: Prebiotic Soda
- Control Group (Active Comparator): Participants will be randomized to continue consumption of traditional non-diet soda.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Prebiotic Soda — Participants will replace traditional non-diet sodas in their diet with a prebiotic soda (OLIPOP). Participants will consume 2 cans/day (24 fl. oz/day) that will add 12 g dietary fiber/day to their diet.
  Arms: Intervention
Behavioral: Active Control — Participants will continue to consume their habitual intake (on average 2-3 servings/day) of traditional non-diet soda.
  Arms: Control Group

SUMMARY:
The main objective of this study is to evaluate the chronic effects of replacing traditional non-diet soda with a prebiotic soda on biomarkers associated with glycemic control in adults with glucose dysregulation who are habitual consumers of traditional soda.

DETAILED DESCRIPTION:
The primary aim of this clinical trial is to evaluate the effects of replacing traditional non-diet soda with a prebiotic soda (i.e., OLIPOP) over an 8 week period on markers of glucose (blood sugar) control in adults with glucose (blood sugar) dysregulation.

Participants (n=224) will be habitual consumers of traditional non-diet sodas, consuming on average 2-3 servings of non-diet soda daily. Participants will be randomized to either an active control group (continued habitual traditional non-diet soda intake, 2 - 3 servings/day) or a behavioral intervention group (OLIPOP prebiotic soda, 2 cans/day, 6 g dietary fiber and 2 - 5 g total sugar per can).

Secondary outcomes will include evaluating the effects of prebiotic soda consumption on additional markers of metabolic health, including long-term glycemic control and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Willing to comply with all study procedures
* Ages 40 - 70 years old
* Habitual consumers of traditional non-diet soda (average intake 2 - 3 servings/daily)
* BMI between 25 - 35 kg/m²
* Waist-to-Hip ratio ≥0.85 for Women and ≥0.9 for Men
* Fasting plasma glucose between 100 - 125 mg/dL
* Consumes ≤16 g total fiber per day to align with the current average dietary fiber intake of American adults
* Non-user or former user (cessation ≥ 12 months) of tobacco or nicotine products
* Non-user of marijuana and hemp products, including CBD products, in the previous 60 days
* Willing to maintain habitual diet (with the exception of study products) and physical activity patterns throughout the trial

Exclusion Criteria:

* Inability to consume a standard 12 fl. oz. carbonated beverage twice daily
* Currently engaged or planning to be on an intensive weight loss regimen program
* Extreme dietary habits or has been diagnosed with an eating disorder
* Habitual use of fiber supplements, inulin-based supplements, acacia fiber, glucomannan, prebiotic supplements, or probiotic supplements within the previous 30 days
* Known allergy or sensitivity to any of the ingredients in the study products
* History or presence of uncontrolled and/or clinically important medical conditions that could interfere with study results interpretation (ex. uncontrolled diabetes mellitus, CKD stage 4-5, severe liver disease/cirrhosis, uncontrolled hypertension, recent myocardial infarction or stroke (within 6 months), severe mental illness or cognitive impairment, immunodeficiency disorders, active infections).
* Gastrointestinal conditions that could potentially interfere with absorption of the study product
* Use of oral or injectable steroids in the previous 90 days
* Use of antibiotic therapy in the previous 90 days
* Unstable use of prescription medications within the previous 90 days that affect plasma glucose levels
* History or presence of cancer, except non-melanoma skin cancer, in the previous 2 years
* Exposure to any non-registered drug product or participation in another intervention study in the previous 30 days
* Recent history (within 12 months) of alcohol or substance abuse
* History of major trauma or surgical event in the previous 60 days
* Person who is pregnant, planning pregnancy, lactating, or unwilling to use contraception during the study period
* Any condition the Investigator believes would interfere with study participation or compliance
* Consumption of pre-biotic sodas in the previous 30 days

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Effects on Fasting Plasma Glucose | Baseline to 8 weeks
  Change in fasting plasma glucose

SECONDARY OUTCOMES:
Effects on Long-term Glycemic Control | Baseline to week 8
  Change in HbA1c
Effect on insulin sensitivity | Baseline to week 8
  Change in fasting plasma insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Lindus Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No